CLINICAL TRIAL: NCT02871791
Title: A Phase 1b/2a Study Of Palbociclib In Combination With Everolimus And Exemestane In Postmenopausal Women With Estrogen Receptor Positive and HER2 Negative Metastatic Breast Cancer
Brief Title: Palbociclib With Everolimus + Exemestane In BC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Sara Tolaney, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-177
Record Dates: First submitted 2016-06-29; First posted 2016-08-18 (Estimated); Results first posted 2022-08-29 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Human Epidermal Growth Factor 2 Negative Carcinoma of Breast; Hormone Receptor (HR)-Positive Breast Cancer
Keywords: Her2-negative metastatic breast cancer; Hormone receptor (HR)-positive breast cancer
MeSH Terms: interventions — palbociclib; Everolimus; exemestane

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Palbociclib, Everolimus, Exemestane (Experimental): * Palbociclib will be administered orally, 100mg, once daily for 21 consecutive days followed by a 7-day rest (28-day cycle)
  * Everolimus will be administered orally, 5mg, once daily on a 28 day schedule
  * Exemestane will be administered orally, 25mg, once daily on a 28 day schedule
  Interventions: Drug: Palbociclib; Drug: Everolimus; Drug: Exemestane

INTERVENTIONS:
Drug: Palbociclib
Drug: Everolimus
Drug: Exemestane

SUMMARY:
This research study is studying a combination of targeted therapy and hormonal therapy as a possible treatment for breast cancer that has spread to other places in the body and is hormone receptor positive (HR+) and HER2-negative.

The names of the study interventions involved in this study are:

* Palbociclib
* Everolimus
* Exemestane

DETAILED DESCRIPTION:
This is a Phase I/II clinical trial. The Phase I portion of this clinical trial tests the safety of an investigational intervention and also tries to define the appropriate dose of the investigational intervention to use for further studies. The Phase II portion of the study tests the safety and effectiveness of an investigational intervention to learn whether the intervention works in treating a specific disease. "Investigational" means that the intervention is being studied.

The FDA (the U.S. Food and Drug Administration) has not approved the combination of Palbociclib, Everolimus, and Exemestane as a treatment for any disease.

This is the first time that the combination of Palbociclib, Everolimus, and Exemestane will be given to humans.

Palbociclib is a drug that may stop cancer cells from growing. Palbociclib blocks activity of two closely related enzymes (proteins that help chemical reactions occur in the body), called Cyclin D Kinases 4 and 6 (CDK 4/6). These proteins are part of a pathway, or a sequence of steps, which is known to regulate cell growth. Laboratory testing has suggested Palbociclib may stop the growth of HR+ breast cancer.

Everolimus is a type of drug called an mTORinhibitor that treats breast cancer by preventing the cells from multiplying by inhibiting the pathway, or a sequence of steps, known to regulate cell reproduction. Everolimus also may stop the growth of cancer cells by decreasing blood supply to the cancer cells.

Exemestane is an anti-hormone therapy that prevents breast cancer cell growth by blocking estrogen receptor stimulation. Premenopausal women will also receive an injection drug called an LHRH (luteinizing hormone-releasing hormone) agonist to shut down ovary function. It is standard of care for people with breast cancer, specifically with HR+ breast cancer, to take anti-hormone therapy.

The combination of everolimus and exemestane is FDA approved to treat this type of breast cancer.

The purpose of the Phase I portion of this research study is to determine a safe and tolerable dose of the combination of Palbociclib, Everolimus, and Exemestane for participants with ER-positive, HER2-negative advanced breast cancer.

The purpose of the Phase II portion of this research study is to determine whether the combination of Palbociclib, Everolimus, and Exemestane is an effective treatment for participants with ER-positive, HER2-negative advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet the following criteria on screening examination to be eligible to participate in the study. Laboratory tests required for eligibility must be completed within 14 days prior to the date of registration. Diagnostic tests, such as MRIs and CT scans, must be performed within 30 days of registration and baseline measurements must be documented within 14 days of the date of registration.
* Participants with histologically or cytologically confirmed hormone receptor (HR)-positive, Her2-negative metastatic breast cancer. Central confirmation of HR positivity is not required
* Postmenopausal women as defined as:

  * Age >60 years

    --- or
  * Age >45 with intact uterus and amenorrhea for ≥ 12 consecutive months or Follicle stimulating hormone (FSH) levels within postmenopausal range according to the ranges established by the testing facility

    --- or
  * Premenopausal women who have been on a GnRH agonist for at least 6 weeks prior to study entry. Women in this group MUST remain on the GnRH agonist for the duration of protocol treatment

    --- or
  * Status post bilateral oophorectomy, after adequate healing post surgery;
* Men are eligible, as long as on a GnRH agonist for at least 6 weeks prior to study entry. Men MUST remain on the GnRH agonist for the duration of protocol treatment.
* Participants must have measurable disease as per RECIST 1.1.
* Prior Treatment Specifics:

  * Participants must have radiological or objective evidence of progression to a CDK4/6 inhibitor regimen in the metastatic setting AND relapse/progression on an NSAI (defined as either relapsed ≤ 12 months after completing adjuvant NSAI or progressed through an NSAI for metastatic or locally advanced breast cancer)
  * Participants may have received any number of previous endocrine/hormonal lines of therapy in the metastatic setting, as long none of them were exemestane-based and the last dose is ≥ 14 days prior to registration;
  * Participants may have received up to one prior chemotherapy line for advanced breast cancer as long as the last dose is ≥ 21 days prior to registration;
  * Participants may have received prior biologic treatments or investigational drugs as long as the last dose is ≥ 21 days prior to registration;
  * Participants may have received radiotherapy for palliative purposes but must not be experiencing > grade 1 treatment related toxicities and have completed treatment ≥ 14 days prior to registration
* Age ≥18 years. Age restriction applies given that no dosing or adverse event data are currently available on the use of palbociclib or exemestane in participants <18 years of age.
* ECOG performance status ≤2 (Karnofsky ≥60%, see Appendix A)
* For participants enrolling the phase IIa part of the study, accessible tumor lesion(s) for the purpose of research biopsy and willingness to undergo a research biopsy before treatment initiation and at the time of disease progression, as well as a single research blood sample before initiation of therapy. Participants who undergo an attempted on-treatment research biopsy and in whom inadequate tissue is obtained are still eligible to receive protocol therapy. They will not be required to undergo a repeat research biopsy attempt.
* For participants enrolling the phase IIa part of the study, willingness to provide archival tumor samples when available.
* Participants must have normal organ and marrow function, as defined below:

  * absolute neutrophil count ≥1,5x109/L
  * platelets ≥100 x109/L
  * total hemoglobin ≥ 9 g/dL (which may be post transfusion)
  * total bilirubin ≤1.5 x institutional upper limit of normal
  * AST(SGOT)/ALT(SGPT) ≤2.5 × institutional upper limit of normal or ≤5 × institutional upper limit of normal for participants with liver metastization
  * creatinine ≤1.5 x above institutional normal or ≥ 60 ml/min/1.73m2 for subjects with creatinine levels above institutional normal.
  * baseline QTc < 500 ms
  * fasting plasma glucose <140 mg/dL / 7.8 mmol/L
* The effects of the combination of palbociclib, everolimus and exemestane on the developing human fetus are unknown. Given that women in this study will be post-menopausal by eligibility criteria (de facto or pharmacologically induced), it is expected that there will be no women of child-bearing potential in this study. If, for any reason, a woman should become pregnant or suspect that she is pregnant while participating in this study, she should inform her treating physician immediately. Of note, premenopausal women and men are only eligible if they have been on a GnRH agonist for at least 6 weeks prior to study entry. These participants MUST remain on the GnRH agonist for the duration of protocol treatment. Such participants should be counseled prior to study entry that GnRH agonists alone may not be adequate contraception and that adequate contraception (barrier method of birth control; abstinence) should be employed for the duration of study participation.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants who have demonstrated intolerance to 125mg of Palbociclib are ineligible for the Phase I portion.
* Participants who are receiving any other investigational agents.
* Participants who have received previous treatment with an mTOR inhibitor or exemestane.
* Participants with a history of allergic reactions attributed to compounds of similar chemical or biologic composition to palbociclib, everolimus or exemestane.
* Participants with known brain metastases may be enrolled in this study if radiation therapy and/or surgery have been completed with a minimum of 3 months of stable disease demonstrated on serial evaluation by CT (with contrast enhancement) or MRI. Such participants must no longer require treatment with corticosteroids or enzyme inducing anti-epileptic medications for their CNS disease.
* Participants with bilateral diffuse lymphangitic carcinomatosis.
* Participants with significant symptomatic deterioration of lung function. If clinically indicated, pulmonary function tests including measures of predicted lung volumes, DLco, O2 saturation at rest on room air should be considered to exclude restrictive pulmonary disease, pneumonitis or pulmonary infiltrates.
* Evidence of current pneumonitis
* Subjects with organ allograft requiring immunosuppression.
* Participants with uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, symptomatic cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements. Ability to comply with study requirements is to be assessed by each investigator at the time of screening for study participation;
  * Impairment of gastrointestinal function or who have gastrointestinal disease that may significantly alter the absorption of study drugs (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea or malabsorption syndrome).
* Participants receiving any medications or substances that are moderate or strong inhibitors or inducers of CYP3A within 7 days of registration. Lists including medications and substances known or with the potential to interact with the CYP3A isoenzymes are provided in Appendix B, and can also be found within Sections 2.4.1.2 and 5.8. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated list such as: http://medicine.iupui.edu/clinpharm/ddis/table.aspx; medical reference texts such as the Physicians' Desk Reference may also provide this information. As part of the enrollment/informed consent procedures, the participant will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the participant is considering a new over-the-counter medicine or herbal product.
* Proton pump inhibitors(PPI) may be taken while on study, however it is recommended that the PPI is taken 12 hours from the time of palbociclib administration. If needed, alternative antacid therapies may be used including H2-receptor antagonists and locally acting antacids. H2-receptor antagonists should be administered with a staggered dosing regimen (twice daily). The dosing of palbociclib should occur at least 10 hours after H2-receptor antagonist evening dose and 2 hours before the H2-receptor antagonist morning dose.
* Pregnant women are excluded.
* Individuals with a history of a different malignancy are ineligible except for the following circumstances: a) if they have been disease-free for at least 5 years and are deemed by the investigator to be at low risk for recurrence of that malignancy; b) if diagnosed with the following cancers and treated within the past 5 years: ductal carcinoma in situ of the breast, cervical cancer in situ, and basal cell or squamous cell carcinoma of the skin.
* Participants known to be HIV-positive on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with palbociclib and everolimus. In addition, these individuals are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in participants receiving combination antiretroviral therapy when indicated. Screening for HIV infection at baseline is not required.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2016-08-24 (Actual); Primary Completion 2020-12-03 (Actual); Study Completion 2021-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sara Tolaney, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: September 12, 2016 to June 26, 2019
Groups:
- Dose 0: Palbociclib 100mg, Everolimus 5mg, Exemestane 25mg: * Palbociclib 100mg will be administered orally, once daily for 21 consecutive days followed by a 7-day rest (28-day cycle)
  * Everolimus 5 mg will be administered orally, once daily on a 28 day schedule
  * Exemestane 25 mg will be administered orally, once daily on a 28 day schedule
- Dose 1: Palbociclib 125mg, Everolimus 5mg, Exemestane 25mg: * Palbociclib 125mg will be administered orally, once daily for 21 consecutive days followed by a 7-day rest (28-day cycle)
  * Everolimus 5 mg will be administered orally, once daily on a 28 day schedule
  * Exemestane 25 mg will be administered orally, once daily on a 28 day schedule
Period: Phase 1b
Arm/Group | Dose 0: Palbociclib 100mg, Everolimus 5mg, Exemestane 25mg | Dose 1: Palbociclib 125mg, Everolimus 5mg, Exemestane 25mg
Started | 6 | 3
Completed | 0 | 0
Not Completed | 6 | 3
Not completed — Death | 0 | 1
Not completed — progressive disease | 6 | 2
Period: Phase 2
Arm/Group | Dose 0: Palbociclib 100mg, Everolimus 5mg, Exemestane 25mg | Dose 1: Palbociclib 125mg, Everolimus 5mg, Exemestane 25mg
Started | 32 | 0
Completed | 29 | 0
Not Completed | 3 | 0
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- [Phase 2a] Palbociclib 100mg, Everolimus 5mg, Exemestane 25mg; [Phase 1b]Dose 0: Palbociclib 100mg, Everolimus 5mg, Exemestane 25mg: * Palbociclib 100 mg will be administered orally, once daily for 21 consecutive days followed by a 7-day rest (28-day cycle)
  * Everolimus 5 mg will be administered orally, once daily on a 28 day schedule
  * Exemestane 25 mg will be administered orally, once daily on a 28 day schedule
- [Phase 1b]Dose 1: Palbociclib 125mg, Everolimus 5mg, Exemestane 25mg: * Palbociclib 125 mg will be administered orally, once daily for 21 consecutive days followed by a 7-day rest (28-day cycle)
  * Everolimus 5 mg will be administered orally, once daily on a 28 day schedule
  * Exemestane 25 mg will be administered orally, once daily on a 28 day schedule
- Total: Total of all reporting groups
Arm/Group | [Phase 2a] Palbociclib 100mg, Everolimus 5mg, Exemestane 25mg | [Phase 1b]Dose 0: Palbociclib 100mg, Everolimus 5mg, Exemestane 25mg | [Phase 1b]Dose 1: Palbociclib 125mg, Everolimus 5mg, Exemestane 25mg | Total
Number analyzed (Participants) | 32 | 6 | 3 | 41
Age, Continuous [Median (Full Range); unit: years] | 55.5 [36 to 73] | 52 [40 to 67] | 68 [48 to 75] | 55.5 [36 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 6 | 3 | 41
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 29 | 6 | 3 | 38
  Black | 2 | 0 | 0 | 2
  Asian | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 32 | 6 | 3 | 0

OUTCOME MEASURES:

1. Primary Outcome: Clinical Benefit Rate (CBR) [Phase 2a]
Description: CBR is defined as the proportion of participants achieving complete response, partial response or stable disease for more than 6 months (CR+PR+SD ≥ 24 weeks) taking as reference the smallest measurements recorded since the treatment started, including the baseline measurements.
Time Frame: Disease evaluations were performed every 8 weeks (within 24 weeks of initiation of study treatment) or every 12 weeks (greater than 24 weeks of initiation of study treatment). Treatment duration has a median of 111 days and maximum of 681 days.
Measure: Count of Participants; unit: Participants
Groups:
- Palbociclib, Everolimus, Exemestane: * Palbociclib 100mg will be administered orally, once daily for 21 consecutive days followed by a 7-day rest (28-day cycle)
  * Everolimus 5 mg will be administered orally, once daily on a 28 day schedule
  * Exemestane 25 mg will be administered orally, once daily on a 28 day schedule
Arm/Group | Palbociclib, Everolimus, Exemestane
Number analyzed (Participants) | 32
Participants | 6

2. Secondary Outcome: Overall Response Rate (ORR) [Phase 2a]
Description: The objective response rate (ORR) was defined as the proportion of participants achieving complete response (CR) or partial response (PR) based on RECIST 1.1 criteria on treatment.
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib, Everolimus, Exemestane
Number analyzed (Participants) | 32
Participants | 0

3. Secondary Outcome: Disease Control Rate (DCR) [Phase 2a]
Description: The DCR defined as the proportion of patient that has CR+PR+SD>=12 weeks. Response will be assessed among participants eligible for the phase IIa part of the study who received at least one dose of the study drugs at the MTD/RP2D and have measurable disease at screening.
Time Frame: as for outcome 1
Population: 2 patients lost follow-up from the study after treatment begins
Measure: Number (95% Confidence Interval); unit: proportion of patients
Arm/Group | Palbociclib, Everolimus, Exemestane
Number analyzed (Participants) | 30
proportion of patients | 0.563 [0.393 to 0.719]

4. Secondary Outcome: Duration of Response (DOR) [Phase 2a]
Description: Response will be assessed among participants eligible for the phase IIa part of the study who received at least one dose of the study drugs at the MTD/RP2D and have measurable disease at screening. DOR defined based on the duration of stable disease.
Time Frame: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Palbociclib, Everolimus, Exemestane
Number analyzed (Participants) | 32
months | 4.24 [3.68 to 7.82]

5. Secondary Outcome: Median Progression Free Survival (PFS) [Phase 2a]
Description: Progression-free survival based on the Kaplan-Meier method is defined as the duration of time from study entry to documented disease progression (PD) or death. Per RECIST 1.1 criteria: progressive disease (PD) is at least a 20% increase in the sum of longest diameter (LD) of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. PD for the evaluation of non-target lesions is the appearance of one or more new lesions and/or unequivocal progression of non-target lesions.
Time Frame: Disease is evaluated and followed-up every 8 weeks, with median of 20.04 months and maximum of 35.64 months.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Palbociclib, Everolimus, Exemestane
Number analyzed (Participants) | 32
months | 3.8 [2 to 5.4]

ADVERSE EVENTS:
Time Frame: Adverse events are evaluated every 8 days each cycle on treatment, and at the end of the therapy. Treatment duration has a median of 111 days and maximum of 681 days.
Description: Serious adverse events (AEs) were defined as events with treatment-attribution of possibly, probably or definitely and grade 3 or higher per CTCAEv4. All remaining events regardless of treatment attribution were classified as Other AEs. Maximum grade toxicity by type for a patient over time was calculated. No further data is available to specify classification of other beyond the general term.
Groups:
- [Phase 2a] Palbociclib 100mg, Everolimus 5mg, Exemestane 25mg: * Palbociclib 100mg will be administered orally, once daily for 21 consecutive days followed by a 7-day rest (28-day cycle)
  * Everolimus 5 mg will be administered orally, once daily on a 28 day schedule
  * Exemestane 25 mg will be administered orally, once daily on a 28 day schedule
Arm/Group | [Phase 2a] Palbociclib 100mg, Everolimus 5mg, Exemestane 25mg | [Phase 1b]Dose 0: Palbociclib 100mg, Everolimus 5mg, Exemestane 25mg | [Phase 1b]Dose 1: Palbociclib 125mg, Everolimus 5mg, Exemestane 25mg
All-Cause Mortality (participants affected / at risk) | 16/32 | 0/6 | 1/3
Serious Adverse Events (participants affected / at risk) | 28/32 | 5/6 | 3/3
Other Adverse Events (participants affected / at risk) | 32/32 | 6/6 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | [Phase 2a] Palbociclib 100mg, Everolimus 5mg, Exemestane 25mg (N=32) | [Phase 1b]Dose 0: Palbociclib 100mg, Everolimus 5mg, Exemestane 25mg (N=6) | [Phase 1b]Dose 1: Palbociclib 125mg, Everolimus 5mg, Exemestane 25mg (N=3)
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0
Alkaline phosphatase increased (Investigations) | 1 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 4 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 5 | 0 | 0
Neutrophil count decreased (Investigations) | 25 | 4 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Platelet count decreased (Investigations) | 3 | 0 | 2
White blood cell decreased (Investigations) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | [Phase 2a] Palbociclib 100mg, Everolimus 5mg, Exemestane 25mg (N=32) | [Phase 1b]Dose 0: Palbociclib 100mg, Everolimus 5mg, Exemestane 25mg (N=6) | [Phase 1b]Dose 1: Palbociclib 125mg, Everolimus 5mg, Exemestane 25mg (N=3)
Abdominal pain (Gastrointestinal disorders) | 4 | 0 | 0
Alanine aminotransferase increased (Investigations) | 7 | 1 | 0
Alkaline phosphatase increased (Investigations) | 3 | 1 | 0
Allergic reaction (Immune system disorders) | 1 | 0 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Anemia (Blood and lymphatic system disorders) | 2 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 8 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 5 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0
Brachial plexopathy (Nervous system disorders) | 1 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 1 | 0 | 0
Chills (General disorders) | 2 | 0 | 0
Constipation (Gastrointestinal disorders) | 3 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 0
Creatinine increased (Investigations) | 0 | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 4 | 0 | 0
Depression (Psychiatric disorders) | 0 | 2 | 0
Diarrhea (Gastrointestinal disorders) | 10 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 4 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Dysgeusia (Nervous system disorders) | 7 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 | 2 | 1
Edema limbs (General disorders) | 1 | 0 | 0
Endocrine disorders - Other, specify (Endocrine disorders) | 1 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 | 1 | 2
Fatigue (General disorders) | 21 | 3 | 2
Fever (General disorders) | 3 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0
Gait disturbance (General disorders) | 1 | 0 | 0
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 8 | 2 | 1
Hemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hot flashes (Vascular disorders) | 1 | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 3 | 2 | 1
Hypertension (Vascular disorders) | 1 | 0 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 3 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 0 | 0
Investigations - Other, specify (Investigations) | 0 | 3 | 0
Jejunal hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Lip pain (Gastrointestinal disorders) | 1 | 0 | 0
Lung infection (Infections and infestations) | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 1 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 31 | 6 | 3
Nausea (Gastrointestinal disorders) | 11 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 28 | 5 | 3
Oral pain (Gastrointestinal disorders) | 1 | 0 | 0
Pain (General disorders) | 3 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 0
Platelet count decreased (Investigations) | 17 | 2 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 10 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 0 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 10 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0
Stomach pain (Gastrointestinal disorders) | 1 | 0 | 0
Tooth infection (Infections and infestations) | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0
Tracheal fistula (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Upper respiratory infection (Infections and infestations) | 4 | 0 | 0
Urinary frequency (Renal and urinary disorders) | 2 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 3 | 0
Vaginal dryness (Reproductive system and breast disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 5 | 0 | 0
Weight loss (Investigations) | 2 | 1 | 0
White blood cell decreased (Investigations) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-18): https://cdn.clinicaltrials.gov/large-docs/91/NCT02871791/Prot_SAP_000.pdf